CLINICAL TRIAL: NCT07176520
Title: AI-Assisted Rehabilitation for Frail Older Adults Discharged From Community Hospitals: A Hybrid Effectiveness-Implementation Trial
Brief Title: AI-Assisted Rehabilitation In Frailty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SingHealth Community Hospitals (Other)
Collaborators: Jurong Community Hospital, Singapore (Unknown)
Responsible Party: Principal Investigator, Ong Chong Yau, Doctor, SingHealth Community Hospitals
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2025-1300
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Frail
Keywords: hybrid effectiveness-implementation study; pragmatic

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Other): Verbal and written discharge summary, advice, and referral to outpatient physiotherapy (if applicable)
  Interventions: Other: usual care only
- AI-assisted rehabilitation (Active Comparator): AI-assisted rehabilitation on top of usual care
  Interventions: Device: AI-assisted rehabilitation

INTERVENTIONS:
Device: AI-assisted rehabilitation — Receives AI-assisted rehabilitation post-discharge at home in addition to usual care
  Arms: AI-assisted rehabilitation
Other: usual care only — Verbal and written discharge summary, advice, and referral to outpatient physiotherapy (if applicable)
  Arms: Usual care

SUMMARY:
This study investigates the effectiveness and implementation of an AI-assisted rehabilitation tool for adults with frailty in the real-world. The main questions it aims to answer are:

Does AI-assisted rehabilitation among frail adults improve patients' physical outcomes? Is there a particular subgroup of frail subjects that will benefit most from AI-assisted rehabilitation?

Researchers will compare AI-assisted rehabilitation to standard practice (advice and QR link for rehabilitation videos to be done at home) to see if AI-assisted rehabilitation improves clinical outcomes compared to standard practice.

Participants will either:

Undergo an AI-assisted rehab with the AI-sensor tool or a standard practice post-discharge from community hospitals for 12 weeks.

Undergo interval assessments of outcomes. Keep a diary of outpatient rehabilitations (if applicable for the subjects).

DETAILED DESCRIPTION:
This is a pragmatic, randomized controlled study on frail patients discharged from three community hospitals in Singapore.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 21years
* Clinical Frailty Score (CFS) 4 to 6 *
* Provided informed consent (for cognitively impaired persons MMSE<18, next-of-kin or proxy to give consent).
* Have access to smartphone/tablet (own or loaned from investigators)/

Exclusion Criteria:

* Medical conditions precluding safe home exercises or severely affect interaction with AI-tool (angina, vision loss, hearing impairment).
* Cognitive impairment (MMSE<18) and no caregiver to assist with use of tool.
* Participation in structured outpatient physiotherapy (>1 times/week), or day rehab programme.

Ages: 21 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Absolute Functional Gain (AFG) | baseline, 3, 6, 9 and 12 weeks.
  AFG= Functional score (at discharge/follow-up points) - functional score (at admission). Functional score is based on Modified Barthel Index (MBI).

SECONDARY OUTCOMES:
Functional outcome: Short Physical Performance Battery (SPBB) | baseline, 3, 6, 9, 12-weeks
  SPBB is a validated and commonly used tool to evaluate physical performance particularly in older adults. It is based on three timed tasks: gait speed (over short distance of 4 metres), balance tests (side-by-side, semi-tandem, and full-tandem), and repetitive chair sit-to-stand (strength and endurance) performance.45 It is an indicator of vulnerability, is associated with readmissions, and predictive of all-cause mortality.

IPD SHARING:
Plan to Share IPD: No
In accordance to my ethical board and institutional requirements.